CLINICAL TRIAL: NCT06543004
Title: Comparison of the Effects of Bio Ceramic and Epoxy Resin-based Sealers on Postoperative Pain After Root Canal Treatment: A Randomized Controlled Trial at Primary Health Care Corporation, Qatar.
Brief Title: Comparison of the Effects of Bio Ceramic and Epoxy Resin-based Sealers on Postoperative Pain After Root Canal Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Primary Health Care Corporation, Qatar (Other Government)
Responsible Party: Principal Investigator, Dareen Azzouz, Consultant Endodontist, Primary Health Care Corporation, Qatar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUHOOTH-D-24-000
Record Dates: First submitted 2024-07-31; First posted 2024-08-07 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Asymptomatic Apical Periodontitis
Keywords: Bioceramic sealer; Resin based sealer
MeSH Terms: interventions — epoxy resin-based root canal sealer

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The control group will be treated by using Resin based sealer during obturation which will be selected at random.
  Interventions: Combination Product: AH plus sealer
- Intervention (Active Comparator): The comparator group will receive Bioceramic sealer during obturation as intervention which will be selected at random.
  Interventions: Combination Product: Bioceramic sealer

INTERVENTIONS:
Combination Product: AH plus sealer — Root canal sealer will be placed inside the root canals during obturation procedure to seal dentine wall and reinforce the remaining tooth tissue.It will be selected randomly to the study samples.
  Arms: Control Group
Combination Product: Bioceramic sealer — Root canal sealer will be placed inside the root canals during obturation procedure to seal dentine wall and reinforce the remaining tooth tissue.It will be selected randomly to the study samples.
  Arms: Intervention

SUMMARY:
This study aims to compare the effect of bio ceramic sealer and resin-based sealer on the intensity and occurrence of post operative pain in single rooted teeth with asymptomatic apical periodontitis.

DETAILED DESCRIPTION:
Root canal sealers are essential for the success of endodontic treatment. Their physical properties, biocompatibility, and interactions with peri-apical tissues directly affect postoperative pain and healing. Endodontic sealers activate trigeminal nociceptors, leading to the release of CGRP (calcitonin gene-related peptide), which causes pain and a neurogenic inflammatory response. Resin-based sealers are widely used in endodontics due to their superior physicochemical properties. However, they have limitations, including the need for a completely dry canal due to their marked hydrophobicity and their initial cytotoxic activity, which cannot be entirely controlled.

Bio-ceramic sealers represent a new generation of endodontic sealers that are favored by many dental professionals due to their small particle size (less than 2 micrometers), non-toxicity, high tissue compatibility, high hydrophilicity, and minimal dimensional changes. Retrospective studies have shown varying outcomes related to postoperative pain after root canal treatment using resin-based or bio-ceramic sealers.

Aim: This study aims to compare the occurrence and intensity of postoperative pain and analgesic intake after root canal treatment using two different types of root canal sealers.

Methods/Design: This study is a binary outcome randomized trial, following the Consolidated Standards of Reporting Trials (CONSORT) guidelines for randomized trials of non-pharmacologic treatment. The study sample will consist of adult patients with a permanent single-rooted tooth diagnosed with asymptomatic apical periodontitis. Participants will be randomly allocated to be treated in the Endodontic clinic of PHCC Qatar with either resin-based sealers (control group) or bio-ceramic sealers (experimental group) to compare postoperative pain after root canal treatment.

Patients will be observed for occurrence of pain or any other complications at 24 hours, 48 hours, and 7 days post-treatment. Postoperative pain will be assessed using a visual analog scale (VAS) at 24 hours, 48 hours, and one week post-treatment.

Differences in the incidence of postoperative pain and the need for an analgesic will be analyzed using the chi-square test. Differences in pain intensity after treatment will be analyzed using the ordinal (linear) chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Permanent single rooted tooth 1-1 configuration and complete root development.
* Requiring root canal treatment.
* Diagnosed with Asymptomatic apical periodontitis, teeth asymptomatic, periapical index will exhibit an apical radiolucency.
* Willing to Participate.

Exclusion Criteria:

* Medically compromised patients.
* Inability to reach working length, complication during treatment.
* Retreatment teeth, multi rooted teeth.
* Periodontological compromised teeth.
* Uncooperative patients.
* Pregnant patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-10-27 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
post operative pain questionnaire | assessed at 24 hours, 48 hours, and 7 days post-treatment.
  The participants of the study groups will be given a questionnaire to record whether they experienced pain following the root canal treatment after applying each type of the study sealers or no, during the Time frame.

SECONDARY OUTCOMES:
Intensity of postoperative pain | assessed at 24 hours, 48 hours, and 7 days post-treatment.
  The patient will be asked to measure Intensity of their postoperative pain using a Visual Analog Scale. It consist of a straight line, usually 10 centimeters in length, with end point defining the extremes of pain. One end of the line represents no pain(usually marked as 0), while the other end represents' worst imaginable pain' (usually marked as 10) participant mark a point on the line that corresponds to their perceived pain intensity. The distance from the 'no pain' end to the mark is then measured and used to quantify the pain level during Time frame.
Analgesic | assessed at 24 hours, 48 hours, and 7 days post-treatment.
  Analgesic intake recorded, The participants of the study will be asked to record any analgesic taken and the number of the tables during the Time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Dareen Azzouz, Principal Investigator — Primary Health care corporation
Locations (1):
- Primary Health Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
A password protected computer system is used to assure secure data storage.Only encrypted systems are used for storing research data on laptops. A locked file cabinet is used to store research related paper forms.Access to study data is limited to only a few members of the study team.Plans are set to destroy all research generated data after 3 years according to PHCC regulations.The study report / publication will show only aggregate results with no identifiers.
  Only deidentified study data is stored. A code number is used instead of the participant's real name on study data and blood/tissue samples.

REFERENCES:
- [Background] Tan HSG, Lim KC, Lui JN, Lai WMC, Yu VSH. Postobturation Pain Associated with Tricalcium Silicate and Resin-based Sealer Techniques: A Randomized Clinical Trial. J Endod. 2021 Feb;47(2):169-177. doi: 10.1016/j.joen.2020.10.013. Epub 2020 Oct 22. PMID 33098889
- [Background] Zamparini F, Lenzi J, Duncan HF, Spinelli A, Gandolfi MG, Prati C. The efficacy of premixed bioceramic sealers versus standard sealers on root canal treatment outcome, extrusion rate and post-obturation pain: A systematic review and meta-analysis. Int Endod J. 2024 Aug;57(8):1021-1042. doi: 10.1111/iej.14069. Epub 2024 Apr 12. PMID 38606520
- [Result] Khandelwal A, Jose J, Teja KV, Palanivelu A. Comparative evaluation of postoperative pain and periapical healing after root canal treatment using three different base endodontic sealers - A randomized control clinical trial. J Clin Exp Dent. 2022 Feb 1;14(2):e144-e152. doi: 10.4317/jced.59034. eCollection 2022 Feb. PMID 35173897
- [Result] Aslan T, Donmez Ozkan H. The effect of two calcium silicate-based and one epoxy resin-based root canal sealer on postoperative pain: a randomized controlled trial. Int Endod J. 2021 Feb;54(2):190-197. doi: 10.1111/iej.13411. Epub 2020 Oct 17. PMID 32929721